CLINICAL TRIAL: NCT07094373
Title: Validation of Diagnostic Codes for Identifying Chlamydial Infections From TriNetX Electronic Health Record Data in the United States
Brief Title: Validation of Chlamydia Diagnostic Codes in TriNetX US EHR Data
Status: Recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: VAV19180; U1111-1322-6372 (Other Grant/Funding Number: WHO ICTRP)
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chlamydial Infections
MeSH Terms: conditions — Chlamydia Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1 (primary objective): Patients aged 14 to 44 years with an ICD-10-CM diagnosis of chlamydia documented in their EHR OR patients with a NAAT result for chlamydia (either positive or negative) during the study period (2016-2024) from the TriNetX USA Network
- Cohort 2 (secondary objective): Patients aged 14 to 44 years with ≥1 ICD-10-CM diagnosis code for chlamydia between 2016 - 2023 in the MarketScan Commercial Claims and Encounters (CCAE) database
- Cohort 3 (secondary objective): Patients aged 14 to 44 years with ≥1 ICD-10-CM diagnosis code for chlamydia or a positive NAAT result for chlamydia between 2016 -2024 in TriNetX Dataworks USA

SUMMARY:
This study is a pharmacoepidemiologic method study based on the secondary use of pre-existing data that examines whether TriNetX, a global health research network encompassing a worldwide electronic health record (EHR), database in the US is an appropriate real-world data (RWD) source for conducting chlamydia-related research to support the chlamydia trachomatis (CT) messenger Ribonucleic acid (mRNA) vaccine program.

There are two primary objectives for this study:

1. To determine the validity of ICD, Tenth Revision, Clinical Modification (ICD-10-CM) diagnostic codes to identify patients with chlamydial infections using TriNetX EHR data in the US
2. To describe screening or diagnostic testing and treatment patterns in patients with chlamydia using TriNetX EHR data in the US

There are also two secondary objectives for this study:

1. To explore the feasibility of developing a modified algorithm for identifying patients with chlamydia applicable for Merative MarketScan Commercial Claims and Encounters (CCAE) database based on the findings from the primary objectives
2. To compare patient characteristics, use of screening or diagnostic testing, and treatment patterns among patients with chlamydia between TriNetX EHR data and the MarketScan CCAE data in the US

ELIGIBILITY:
Inclusion Criteria for Primary Objectives:

* Patients with an ICD-10-CM diagnosis of chlamydia documented in their EHR OR patients with a nucleic acid amplification test (NAAT) result for chlamydia (either positive or negative) during the study period. The index date is the date of the first-recorded diagnosis code, or the date of the first-recorded NAAT result when no diagnosis code for chlamydia exists.
* Patients with at least one visit within 30 days both before and after their index date.

Exclusion Criteria for Primary Objectives:

* Patients with no documented ICD-10-CM diagnosis for chlamydia who possessed unknown laboratory test results for chlamydia during the study period (removed from ICD validation assessment in primary analysis).
* Patients with an ICD-10-CM diagnosis without a corresponding laboratory test (removed from ICD validation assessment in primary analysis).

Note: The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 14 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: For the primary objectives, the study population will include patients aged 14 to 44 years old identified between 1 January 2016 and 31 October 2024 in TriNetX USA Network. Patients are eligible if they have at least one ICD-10-CM diagnosis code for chlamydia or a known Nucleic Acid Amplification Test (NAAT) result.
  For the secondary objectives, the study population includes 1.) patients aged 14 to 44 years with at least one ICD-10-CM diagnosis code for chlamydia between 1 February 2016 and 30 November 2023 in the MarketScan CCAE database and 2.) patients aged 14 to 44 years with an ICD-10-CM diagnosis code for chlamydia or a positive NAAT result for chlamydia between 1 January 2016 and 31 October 2024 in TriNetX Dataworks USA.
Sampling Method: Non-Probability Sample
Enrollment: 533000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Validity of ICD-10-CM Diagnostic Codes for Chlamydial Infections | From year 2016 through year 2024
  Diagnostic performance of ICD-10-CM codes for chlamydial infections, including sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV), compared to Nucleic Acid Amplification Test (NAAT) results for chlamydial infections
Descriptive analyses of chlamydia patients | From year 2016 through year 2024
  Describe demographic characteristics, laboratory testing, and treatment patterns among true positive and false negative chlamydia patients

SECONDARY OUTCOMES:
Validity of CCAE Database for Chlamydial Infections | From year 2016 through year 2023
  Detect chlamydia cases using a mix of diagnostic codes, lab test codes, treatments, to detect/confirm chlamydia infection
Comparison of chlamydia patient characteristics between EHR and claims RWD sources in the US | From year 2016 through year 2024
  Compare demographics and clinical features (e.g., age, sex, treatment history, comorbidities) of chlamydia patients as seen in EHRs which contain clinical notes, lab results, and detailed medical histories and claims data

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org